CLINICAL TRIAL: NCT00607763
Title: A Phase 1, Open-Label Study Of The Safety And Pharmacokinetics Of Repeated-Dose Micafungin (FK463) In Infants And Toddlers (≥4 Months TO < 24 Months Of Age) With Esophageal Candidiasis Or Other Invasive Candidiasis
Brief Title: Study of Mycamine® in Infants and Toddlers With Fungal Infections to Evaluate Safety and Blood Levels of the Drug
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: 9463-CL-2102
Record Dates: First submitted 2008-01-23; First posted 2008-02-06 (Estimated); Last update posted 2014-08-20 (Estimated); Status verified 2014-08

CONDITIONS: Invasive Candidiasis; Esophageal Candidiasis; Oropharyngeal Candidiasis; Candidemia
Keywords: Antifungal; Echinocandin; Candidiasis; Micafungin
MeSH Terms: conditions — Candidiasis, Invasive; Candidemia; Candidiasis | interventions — Micafungin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1. Micafungin (Experimental)
  Interventions: Drug: Micafungin (Mycamine)

INTERVENTIONS:
Drug: Micafungin (Mycamine) — IV
  Other Names: FK463

SUMMARY:
Infants and toddlers with fungal infections will receive 10 to 14 days of treatment with an antifungal drug. Safety and drug blood levels will be assessed

DETAILED DESCRIPTION:
This is a prospective, multicenter, open-label, repeat-dose study. Subjects will receive treatment with intravenous micafungin for 10 to 14 days (per investigator clinical judgment) at a daily dose of 4.5 mg/kg (determined by the subject's weight at baseline). Serial blood samples for assessment of pharmacokinetics will be collected.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is ≥4 months to < 24 months
2. Subject has suspected, proven or probable candidiasis, candidemia or other invasive candidiasis
3. Subject has sufficient venous access to permit administration of study medication, collection of pharmacokinetic samples, and monitoring of laboratory safety variables

Exclusion Criteria:

1. Subject has evidence of significant liver disease, as defined by aspartate transaminase (AST), alanine transaminase (ALT), bilirubin or alkaline phosphatase > 5 times the upper limit of normal (ULN)
2. Subject has a concomitant medical condition that in the opinion of the investigator and/or medical monitor precludes enrollment into the study
3. Subject has a history of anaphylaxis, hypersensitivity, or any serious reaction to the echinocandin class of antifungals
4. Subject has received treatment with an echinocandin within one week prior to first dosing
5. Subject status is unstable and subject is unlikely to complete all study required procedures

Ages: 4 Months to 23 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 9 (Actual)
Dates: Start 2007-10; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Evaluation of Micafungin pharmacokinetics | 10 - 14 Days

SECONDARY OUTCOMES:
Assess safety and tolerability of micafungin by adverse events, vital signs, hematology and chemistry laboratory tests, ECGs and physical evaluation | Day 1 to End of Study

CONTACTS AND LOCATIONS:
Overall Officials: Central Contact, Study Director — Astellas Pharma Global Development
Locations (6):
- United States (6):
  - Los Angeles, California
  - Orange, California
  - Louisville, Kentucky
  - Kansas City, Missouri
  - Dallas, Texas
  - Houston, Texas